CLINICAL TRIAL: NCT01931397
Title: Novel Use of Dried Blood Spots (DBS)for Home Monitoring in Children With Kidney
Brief Title: DBS for Home Monitoring in Children With Kidney Transplantation
Acronym: DBS
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Amira Al-Uzri, Professor of Pediatrics, Oregon Health and Science University
Other Study IDs: PROG-12G03
Record Dates: First submitted 2013-08-16; First posted 2013-08-29 (Estimated); Results first posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Kidney Disease
Keywords: Dried blood spots; kidney transplant; Children
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Kidney transplantation is the treatment of choice for kidney failure in children. Kidney transplant recipients need to take immunosuppression for the rest of their lives after transplantation to prevent rejection of the graft. One of the important medications is called Tacrolimus which can prevent rejection of the kidney graft but at the same time is toxic to the kidney. Therefore, repeated blood levels of Tacrolimus with tests of kidney function will help physicians to prescribe the best dose for therapy to prevent kidney rejection and kidney toxicity. Failure of compliance with taking Tacrolimus is also an important cause of graft failure especially among teenagers, so repeated blood Tacrolimus levels are necessary to detect patients who fail to take their medications on a regular basis. We have developed a lab assay that measures Tacrolimus blood level and creatinine (for kidney function) using one dried blood spot (DBS) on filter paper similar to the filter paper used in the new born screen. We plan to teach patients how to do the test at home once a month and mail the filter paper back to OHSU for analysis for Tacrolimus and creatinine. The advantage of this method is that it is less painful for children then a regular blood dray from the vein, can be done easily at home, will be most cost effective as it will save the family a day of work or school and can detect both the Tacrolimus level and the kidney function at the same time.

We will assess the effect of doing this simple finger prick at home on compliance, on Tacrolimus levels and kidney function over the study period of one year. We will also assess how satisfied patients are with this method instead of going to the lab or the hospital for blood test. All subjects will continue on their regular clinic visits and will continue to have their routine blood draws by intravenous method in the lab during the study.

DETAILED DESCRIPTION:
Specific Aim 1: To validate the DBS method as a home monitoring device for use at home by parents and patients in 30 pediatric kidney transplant recipients. We will validate the TAC and creatinine (Cr) blood levels obtained by DBS method in comparison to blood TAC and serum creatinine levels using standard laboratory assays in CLIA approved clinical laboratories.

Specific Aim 2: The use of DBS on filter papers is associated with better adherence to monthly blood testing and medication intake. This aim can be tested by assessing the number of DBS on filter papers that are returned to OHSU every month. Adherence with medication intake will be assessed by measuring the variability of TAC trough levels, and by individual reporting.

We will calculate the percent of returned DBS filter papers to OHSU on a monthly basis as well as the percent of those that are collected properly at home and are successfully utilized for TAC and Cr analysis.

Specific Aim 3: This aim will explore patient and family satisfaction and self management using DBS method vs. the standard method of scheduled clinic and laboratory visits.

Design: This is a pilot study to evaluate and validate the novel use of DBS on filter paper as a home monitoring method. This study will involve within-subjects, repeated measures design to test specific hypotheses.

Participants: The pediatric kidney transplant program at Doernbecher Children's Hospital/OHSU follows approximately 120 active renal transplant recipients between 2-21 years. Thirty patients of both genders will participate in this study and will be followed for one year.

Inclusion criteria:

1. On Tacrolimus immunosuppression therapy
2. At least six months post kidney transplantation

ELIGIBILITY:
Inclusion Criteria:

Kidney transplant recipients between the ages of 2-21 years at time of enrollment

1. On Tacrolimus immunosuppression therapy
2. At least six months post kidney transplantation

Exclusion Criteria:

Not on tacrolimus therapy Less than 6 months after kidney transplantation Refusal to provide consent fomr

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children who are followed at the Pediatric Kidney Transplant CLinic at OHSU.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amira Al-Uzri, MD, MCR, Principal Investigator — Oregon Health and Science University
Locations (1):
- Doernbecher Children's Hospital /OHSU, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Cohort: This is a prospective non randomized study. All patients were approached at the pediatric kidney transplant clinic at OHSU in a non randomized fashion until the target enrollment of 30 patients was met.
Period: Overall Study
Arm/Group | Total Cohort
Started | 30
Completed | 19
Not Completed | 11
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 8
Not completed — moved out of state | 1

BASELINE CHARACTERISTICS:
Population: Descriptive
Arm/Group | Total Cohort
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — Age (years) at time of enrollment
  years | 13.6 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Number of years post kidney transplantation [Mean (Standard Deviation); unit: years] | 5.93 (4.57)

OUTCOME MEASURES:

1. Primary Outcome: Variability of Tacrolimus Blood Levels Measured by DBS Over Time
Description: Mean standard deviation scores for Tacrolimus blood levels obtained by DBS for each patient over time.
Time Frame: 12 months
Population: 9 participants were excluded from final analysis because they submitted two or less evaluable blood samples. A total of 216 DBS samples were received during the study
Measure: Mean (Standard Deviation); unit: ng/ml
Units Other Than Participants: blood samples
Arm/Group | Total Cohort
Number analyzed (Participants) | 21
Number analyzed (blood samples) | 216
ng/ml | 2.635 (1.086)

2. Secondary Outcome: Percentage of Families Preferring DBS Method
Description: The % of families who anticipated preference of DBS method over intravenous blood draws at the time of enrollment and then the % of those who preferred DBS at end of study period (12 months).
  Families include parents/caregivers and participants who are over 10 years of age were asked to fill in the preference scale separately.
  Preference for DBS Testing was measured using a Visual Analog Scale (VAS) on which a zero was equivalent to no preference for DBS versus laboratory-based monitoring and on which positive numbers indicated greater preference for DBS (up to +72) and negative scores indicated a greater preference for laboratory-based monitoring (down to -72).
Time Frame: At baseline and then at 12 months
Population: 25 families participated in the preference survey at time of enrollment and only 15 families completed the survey at the end of the study period (12 months).
Measure: Number; unit: % of families
Groups:
- At Time of Enrollment: Number of families at enrollment
- At End of Study: Numbers of families at end of study
Arm/Group | At Time of Enrollment | At End of Study
Number analyzed (Participants) | 25 | 15
% of families | 88 | 93

3. Other Pre Specified Outcome: Mean Tacrolimus Blood Levels Measured by DBS Over Study Period According to Age
Description: Mean Tacrolimus blood levels obtained by DBS in each patient over their time in the study in children who are 12 years and over versus those less than 12 years of age.
Time Frame: up to 12 months
Population: We analyzed a total of 216 dried blood spots for Tacrolimus blood levels measured in ng/ml
Measure: Mean (Standard Deviation); unit: ng/ml
Units Other Than Participants: number of blood samples
Groups:
- Group 1: Participants 12 years and over
- Group 2: Participants less than 12 years of age
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 21 | 9
Number analyzed (number of blood samples) | 126 | 90
ng/ml | 2.73 (1.21) | 2.81 (1.16)

4. Other Pre Specified Outcome: Changes in Adherence Parameters to Home DBS Method
Description: We will calculate the percent of returned DBS filter papers to OHSU on a monthly basis utilized for TAC and Cr analysis.
  we calculated the percentage as the number of DBS that were actually received divided by the total number of DBS expected to be received from participants over the study time period
Time Frame: At baseline then every 3 months for 12 months
Population: The number of DBS cards expected to be received by those 28 patients were 279 DBS samples.
Measure: Number; unit: percentage of DBS cards
Units Other Than Participants: Total number of DBS cards
Arm/Group | Total Cohort
Number analyzed (Participants) | 28
Number analyzed (Total number of DBS cards) | 279
percentage of DBS cards | 77

ADVERSE EVENTS:
Arm/Group | Total Cohort
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
This is a pilot study to assess the feasibility of doing home dried blood spot sampling.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No